CLINICAL TRIAL: NCT02210611
Title: 36 Versus 42 Hour Time Interval From Ovulation Induction to Intrauterine Insemination in Stimulated Cycles With GnRH Antagonists
Brief Title: 36 Versus 42 Hour Time Interval From Ovulation to Intrauterine Insemination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruition too slow
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0038-14-EMC
Record Dates: First submitted 2014-07-30; First posted 2014-08-07 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 36 hours (Active Comparator): Intrauterine insemination 36 hours after ovulation induction
  Interventions: Procedure: Intrauterine Insemination 36 hours
- 42 hours (Active Comparator): Intrauterine insemination 42 hours after ovulation induction
  Interventions: Procedure: Intrauterine Insemination 42 hours

INTERVENTIONS:
Procedure: Intrauterine Insemination 36 hours — Intrauterine insemination 36 hours after ovulation induction
  Arms: 36 hours
Procedure: Intrauterine Insemination 42 hours — Intrauterine insemination 42 hours after ovulation induction
  Arms: 42 hours

SUMMARY:
The purpose of this study is to prove that a higher clinical pregnancy rate can be achieved with a 42 to 44 hour time interval between ovulation trigger and intrauterine insemination than a 36 to 38 hour time interval in stimulated cycles utilizing gonadotropins and GnRH antagonists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can be monitored for follicle growth and hormone measurements on the day of ovulation trigger, or one day before.
2. Patients who have no more than 4 follicles of 14 mm or more
3. Patients who have no more than 6 follicles of 10 mm or more

Exclusion Criteria:

1. Patients who cannot give informed consent to language or comprehension barriers
2. Patients who are deemed to be at high risk for high order multiple gestations
3. Patients who cannot be monitored on the day of hCG administration or one day before

Ages: 17 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks following insemination

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weiss, MD, Principal Investigator — Haemek Medical Center, Afula, Israel
Locations (1):
- Emek Medical Center, Afula, Israel